CLINICAL TRIAL: NCT00674141
Title: Nasal Administration of Dexamethasone for MS Treatment
Brief Title: Nasal Administration of Dexamethasone for Multiple Sclerosis (MS) Treatment
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: was not approved by the ministry of health
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Dminitrios Karussis, Hadassah Medical Organization
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS089-HMO-CTIL
Record Dates: First submitted 2008-05-06; First posted 2008-05-07 (Estimated); Last update posted 2010-06-03 (Estimated); Status verified 2008-05

CONDITIONS: MS Patient With Relpasing Remitting Attacks
Keywords: Multiple Sclerosis, relapsing remitting, Dexamethasone
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): only one experimental treated group
  Interventions: Drug: Dexamethasone soduim phosphate

INTERVENTIONS:
Drug: Dexamethasone soduim phosphate — nasale administation of Dexamethasone in 20mg dose/day (in two divided doses) fpr sevem days of treatment

SUMMARY:
The study aims to assess the safety and efficacy of nasale administration of Dexamethasone in relapsing MS patients

ELIGIBILITY:
Inclusion Criteria:

* MS patients with esatblished relapsing remitting attacks
* increase in EDSS of at least 1 point for a least one day

Exclusion Criteria:

* children under 18
* pregnant patients
* patients with diabetes
* known allergy to steroids
* patients who received steroids within 3 months prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-12 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
reduction in the EDSS functional system score | four months

CONTACTS AND LOCATIONS:
Overall Officials: Elka Touitou, PhD, Prof., Principal Investigator — Hebrew University, Jerusalem. Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel